CLINICAL TRIAL: NCT03142542
Title: A Randomized, Double-blind, Placebo-controlled, Investigator Initiated Clinical Trial to Evaluate the Efficacy and Safety of Udenafil Dosed Once a Day in Patients With Erectile Dysfunction After Bilateral Nerve-sparing Radical Prostatectomy
Brief Title: The Efficacy and Safety of Udenafil in Patients With Erectile Dysfunction After Bilateral Nerve-sparing Radical Prostatectomy
Acronym: DA8159_EDP_IIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seong Soo Jeon, Principal Investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-02-112
Record Dates: First submitted 2017-04-11; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer With Radical Prostatectomy

STUDY DESIGN:
Intervention Model Description: placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Udenafil 75mg (Experimental): Drug: Udenafil 75mg by mouth, once daily, for 32 weeks
  Interventions: Drug: ZYDENA TAB.75mg(Udenafil 75mg)
- Placebo (Placebo Comparator): Drug: placebo by mouth, once daily, for 32 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ZYDENA TAB.75mg(Udenafil 75mg) — ZYDENA TAB.75mg(Udenafil 75mg): by mouth, Once daily, for 32 weeks
  Arms: Udenafil 75mg
Drug: Placebo Oral Tablet — Placebo Oral Tablet: by mouth, Once daily, for 32 weeks
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of Udenafil dosed once a day in patients with erectile dysfunction after bilateral nerve-sparing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 20 or over 20 years and not more than 70 years who underwent bilateral nerve-sparing radical prostatectomy due to prostate cancer without metastasis
* IIEF-EF score ≥22 at 1-8 weeks before bilateral nerve-sparing radical prostatectomy, and IIEF-EF ≤16 at screening visit
* Presence of sexual partner from 8 weeks before bilateral nerve-sparing radical prostatectomy, and had planned to keep it during the trial
* Agreed not to use any other erectile dysfunction medication (including both generic and specialty medicines) and other erectile dysfunction therapies during the trial period.
* Patient agrees to voluntary participation and follow the instructions carefully, after fully hearing and understanding the details of this clinical trial

Exclusion Criteria:

* Patient who needs additional treatment in addition to bilateral nerve- sparing radical prostatectomy
* Use Inhibitors of PDE-5 (Viagra®, Levitra®, Cialis®, Zydena®, Yaila®, Mvix® and Generic Medicines) or autologous injections of vasodilators or other erectile dysfunction therapies for erectile dysfunction within the first 8 weeks of bilateral nerve-sparing radical prostatectomy
* If there is an uncontrolled diabetes (HbA1C> 12%) at Visit 1
* If there is proliferative diabetic retinopathy at Visit 1
* If there is a history of CABG surgery, stroke, unstable angina, myocardial infarction, life-threatening arrhythmia, or heart failure within 6 months before the screening visit
* History of spinal cord injury, non nerve-sparing radical prostatectomy or radical pelvic surgery
* Hypotension below 90 / 50mmHg or uncontrolled hypertension above 170 / 100mmHg
* Penis anatomic abnormalities (severe penile fibrosis, Peyronie's disease, etc.)
* Presence of serious disability such as malignant tumor, lung, blood, endocrine system in Visit 1
* Patient who have active hepatitis B or C or who are infected with HIV virus
* Patient who have genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency, glucose-galactose uptake disorder
* Patient who have hyperprolactinemia or hypothyroidism

  * Serum AST and ALT are three times higher than normal upper limit
  * Serum Creatinine ≥ 2.5 mg / dl
* Patient who have retinitis pigmentosa
* Patient who have blood disease (sickle cell disease, multiple myeloma, leukemia) or bleeding disorder that can cause priapism
* Patient with congenital QT prolongation syndrome or those taking a drug that increases QT interval
* If the examiner considers that he / she is not suitable for participation in clinical trials, such as mental disorder or persistent abuse of medication
* Patient who is taking Nitrate / Nitric oxide (NO) donor (Nitroglycerin, Sodium nitroprusside, Isosorbide mononitrate / dinitrate, Amyl nitrate / nitrite, etc.)
* Patient who is taking Guanylate Cyclase stimulator (such as Riociguat)
* Patient who is taking warfarin
* Patient who is taking medications or foods that affect CYP3A4 metabolism

  * Metabolic inhibitors: Antibacterials (Erythromycin, etc.), Antifungals (Itraconazole, etc.), Antivirals (Ritonavir, Saquinavir, Amprenavir, Indinavir, Nelfinavir, etc.), H2 receptor antagonist (Cimetidine, etc), or grapefruit juice
  * Metabolic inducers: Dexamethasone, Rifampicin, Antipyretics (Phenytoin, Phenobarbital, Carbamazepine, etc.)
* Patient who is taking androgens (Testosterone, etc.) or anti-androgens (5α-reductase inhibitors such as Finasteride, Dutasteride and anti- androgen hormones such as Flutamide and Bicalutamide)
* Patient who is taking Trazodone
* Patient who received other clinical trial medications (including placebo) within 4 weeks before the screening visit
* History of hypersensitivity reactions to PDE-5 inhibitors (Viagra®, Levitra®, Cialis®, Zydena®, Yaila®, Mvix® and each Generic drug)
* Patient who did not respond to PDE-5 inhibitors (Viagra®, Levitra®, Cialis®, Zydena®, Yaila®, Mvix® and each Generic drug)
* Patient who has hypoactive sexual desire
* If the examiner judges that it is not suitable for participation in this trial

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who has IIEF-EF score ≥22 | at 32 weeks
  The IIEF-EF score is International Index of Erectile Function - Erectile Function. The Questionaire is composed of 6 questions.

SECONDARY OUTCOMES:
Safety evaulation: Occurrence of any adverse events | for 32 weeks
  The AE is evaluated for grade, intensity, relationship by protocol definition
Safety evaluation: Systolic and diastolic blood pressure | for 32 weeks
  by Physical exam, mmHg
Safety evaluation: 12-lead ECG | for 32 weeks
  ECG test
Safety evaluation: Number of Participants With Abnormal Laboratory Values | for 32 weeks
  Blood and urine test
Safety evaluation:pulse rate | for 32 weeks
  by Physical exam, beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: SeongSoo Jeon, PhD, Principal Investigator — Samsung Medical Center